CLINICAL TRIAL: NCT01167894
Title: A Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover Bioequivalence Study of Simvastatin 80 mg Tablets of Dr. Reddy's to be Compared With Zocor® 80 mg Tablets of Merck & Co. Inc., USA in Healthy Adult Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Simvastatin Tablets 80 mg of Dr. Reddy's Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. M.S. Mohan / Vice President (Research and Development), Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8331
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Simvastatin
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Experimental): Simvastatin 80 mg tablets Dr. Reddy's Laboratories Ltd.
  Interventions: Drug: Simvastatin
- Zocor (Active Comparator): Zocor® 80 mg tablets of Merck & Co. Inc., USA
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 80 mg tablets Dr. Reddy's Laboratories Ltd
  Other Names: Zocor® 80 mg tabletsof Merck & Co. Inc., USA

SUMMARY:
The purpose of this study is to

* compare the single dose bioavailability of Simvastatin 80 mg tablets with Zocor® 80 mg tablets of MercK & Co. Inc, USA in healthy subjects under fasting conditions
* monitor adverse events and to ensure the safety of subjects.

DETAILED DESCRIPTION:
A randomized, two-treatment, two-period, two-sequence, single dose, crossover bioequivalence study of Simvastatin 80mg tablets of Dr. Reddy's Laboratories Limited to be compared with Zocor® 80 mg tablets of Merck & Co. Inc., USA in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will provide written informed consent.
* Subjects must be healthy adults within 18-45 years of age (inclusive) weighing at least 50 kg.
* Subjects must be within ±10% of ideal body weight in relation to height according to Life Insurance Corporation of India height-weight chart for non-medical cases.
* Subjects must be of normal health as determined by medical history and physical examination performed within 15 days prior' to the commencement of the study.
* Have normal ECG, X-ray and vital signs.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.
* If subject is a female volunteer and

  * is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device, or abstinence.
  * is postmenopausal for at least 1 year.
  * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject) No female volunteers turned up to the site for participating in the study.

Exclusion Criteria:

Bioequivalence studies are usually conducted in healthy adult subjects in order to assess and compare the pharmacokinetic profile of test and reference formulations under uniform conditions. Therefore it is essential to exclude those subjects who show abnormalities with respect to their health parameters. Subjects were excluded to participate in the study based on certain criteria. These criteria were made in order to safeguard the health of the subjects enrolled into the study.

* Subjects incapable of understanding the informed consent.
* Subjects with BP≤90/60 or BP≥140/90
* History of hypersensitivity or idiosyncratic reaction to Simvastatin.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal, endocrine, immunologic, neurologic and haematologic function.
* Regular smoker who smokes more than ten cigarettes daily and has difficulty in abstaining from smoking for the duration of each study period.
* Subjects who has taken over the counter or prescribed medications, including any enzyme modifying drugs or any systemic medication within the past 30 days prior to start of clinical period.
* History of any psychiatric illness, which may impair the ability to provide written, informed consent.
* Subjects who have a history of alcohol or substance abuse within the last 5 years.
* Subjects with clinically significant abnormal values of laboratory parameters.
* Subjects who have participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 3 months.
* Subjects who tested positive at screening for Human Immunodeficiency Virus, Hepatitis B Surface Antigen or Hepatitis C Virus
* Subjects with positive urine screen for drugs of abuse.
* Any subject in whom Simvastatin is contraindicated for medical reasons.
* Subjects who have used any drugs or substances such as herbal preparations known to be strong inhibitors of CYP.enzymes (formerly known as cytochrome P450 enzymes) within 14 days prior to the first dose.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are-currently breast-feeding. No female volunteers reported to study site for participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2005-01; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mangesh Kulkarni, Principal Investigator — Vimta Labs Limited, Hyderabad, India, 500 051